CLINICAL TRIAL: NCT02288676
Title: DOvEEgene/WISE Genomics: Diagnosing Ovarian and Endometrial Cancer Early Using Genomics
Acronym: DOvEEgene
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Lucy Gilbert, Professor, Department of Obstetrics and Gynecology & Department of Oncology, McGill University
Other Study IDs: A08-M79-13B
Record Dates: First submitted 2014-10-28; First posted 2014-11-11 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Neoplasms; Endometrial Neoplasms; Endometrial Cancer; Ovarian Cancer; Screening; Safety; Reduced Mortality; Reduced Morbidity; Early Diagnosis
Keywords: genomics; somatic mutations; genetic mutations; high-grade serous cancer; ovarian cancer; endometrial cancer; DNA tagging
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Case Group: Participants must have suspected or confirmed upper genital tract cancer (uterine, tubal and ovarian) and must be scheduled to undergo surgery for tumor removal.
- Control Group: Participants must not be under investigation for any pre-cancerous or cancerous lesions of the genital tract, and must be scheduled for a hysterectomy, bilateral salpingectomy with/without bilateral oopherectomy for presumed benign condition.

SUMMARY:
This study aims to develop and validate a test for detecting ovarian and endometrial cancers early. It relies on detecting somatic mutations that are associated with these cancers from a uterine pap test. A saliva sample is also collected that acts as an internal control and has the ability to detect deleterious germline mutations associated with common hereditary cancers (such as breast, ovarian, endometrial, colon, and pancreatic cancers). A machine learning classifier is then used to discriminate between cancer and benign disease.

DETAILED DESCRIPTION:
For women in high-income countries, ovarian/fallopian tube and endometrial cancers are within the top four cancers in terms of incidence, death and healthcare expenditure. The deaths associated with these cancers are largely caused by Stage III/IV disease, for which cure rates have not changed in three decades, despite escalating costs of treatment. Attempts at early detection have been ineffective in reducing mortality, because the high-grade subtypes, which account for the majority of deaths, metastasize while the primary cancer is still small, has not caused symptoms, and is undetectable by imaging or blood tumour markers.

In recent years, the recognition that somatic mutations are early steps in carcinogenesis has led to a shift from tests such as imaging and non-specific blood tumour markers to technology that detects cancer-associated mutations in cervical, uterine, or blood samples. Several DNA-tagging technologies have been shown to be capable of identifying small amount of cancer DNA among thousands of normal cells, the proverbial needle in a haystack.

This investigation aims to develop and validate a high-sensitivity capture using a panel of genes involved in ovarian and endometrial carcinogenesis, low-pass whole genome sequencing, coupled with a machine-learning derived classifier for discriminating cancer from benign gynecologic disease prevalent in peri/post-menopausal women.

ELIGIBILITY:
Case Inclusion:

* Subjects should have suspected or confirmed cancer of the upper genital tract.
* Participant will undergo surgery for tumour removal.

Control inclusion:

• Subjects should be scheduled to have a hysterectomy, bilateral salpingectomy, with or without bilateral oophorectomy, for presumed benign disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participating hospitals run multiple weekly routine gynecology and gynecologic oncology clinics. The cases include women scheduled to undergo surgery for tumor removal, for either proven or suspected upper genital tract cancer. The controls include women scheduled to have a hysterectomy, bilateral salpingectomy (removal of the fallopian tubes) with/without bilateral oophorectomy (removal of the ovaries) to treat benign conditions.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Detection of cancer-related mutations | 3 years
  Diagnosis ovarian and endometrial cancers by detection of cancer-related mutation taken by brush sample of uterus with high sensitivity and specificity.

SECONDARY OUTCOMES:
Patient related outcomes including pain and acceptability | 3 years
  Pain scores reported by participants on numeric pain and discomfort scale (NPS). Patients' attitude towards the test including willingness to have it done on an annual basis will be evaluated.
Risks associated with the DOvEEgene test | 3 years
  Evaluate all risks associated with the DOvEEgene test including complications from the sampling technique as well as unnecessarily interventions resulting from false positive tests.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ioannis Ragoussis, PhD, Study Director — McGill Genome Center
Locations (1):
- Royal Victoria Hospital (Glen Site), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilbert L, Basso O, Sampalis J, Karp I, Martins C, Feng J, Piedimonte S, Quintal L, Ramanakumar AV, Takefman J, Grigorie MS, Artho G, Krishnamurthy S; DOvE Study Group. Assessment of symptomatic women for early diagnosis of ovarian cancer: results from the prospective DOvE pilot project. Lancet Oncol. 2012 Mar;13(3):285-91. doi: 10.1016/S1470-2045(11)70333-3. Epub 2012 Jan 17. PMID 22257524
- [Background] Kinde I, Bettegowda C, Wang Y, Wu J, Agrawal N, Shih IeM, Kurman R, Dao F, Levine DA, Giuntoli R, Roden R, Eshleman JR, Carvalho JP, Marie SK, Papadopoulos N, Kinzler KW, Vogelstein B, Diaz LA Jr. Evaluation of DNA from the Papanicolaou test to detect ovarian and endometrial cancers. Sci Transl Med. 2013 Jan 9;5(167):167ra4. doi: 10.1126/scitranslmed.3004952. PMID 23303603
- [Background] Gilbert L, Revil T, Meunier C, Jardon K, Zeng X, Martins C, Arseneau J, Fu L, North K, Schiavi A, Ehrensperger E, Artho G, Lee T, Morris D, Ragoussis J. The empress of subterfuge: cancer of the fallopian tube presenting with malapropism. Lancet. 2017 Sep 2;390(10098):1003-1004. doi: 10.1016/S0140-6736(17)31586-6. No abstract available. PMID 28872014
- [Background] Wang Y, Li L, Douville C, Cohen JD, Yen TT, Kinde I, Sundfelt K, Kjaer SK, Hruban RH, Shih IM, Wang TL, Kurman RJ, Springer S, Ptak J, Popoli M, Schaefer J, Silliman N, Dobbyn L, Tanner EJ, Angarita A, Lycke M, Jochumsen K, Afsari B, Danilova L, Levine DA, Jardon K, Zeng X, Arseneau J, Fu L, Diaz LA Jr, Karchin R, Tomasetti C, Kinzler KW, Vogelstein B, Fader AN, Gilbert L, Papadopoulos N. Evaluation of liquid from the Papanicolaou test and other liquid biopsies for the detection of endometrial and ovarian cancers. Sci Transl Med. 2018 Mar 21;10(433):eaap8793. doi: 10.1126/scitranslmed.aap8793. PMID 29563323